CLINICAL TRIAL: NCT04626193
Title: Comparing the Efficacy of Two Weeks Therapy of Doxycycline,Levofloxacin,Tinidazole Versus Levofloxacin With Tinidazole on Rate of Eradication of Helicobacter Pylori Infected Patients on Syrian Population
Brief Title: LOAD VS Levofloxacine Concomitant
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Damascus Hospital (Other)
Responsible Party: Principal Investigator, Marouf Alhalabi, head of digestive diseases department, Damascus Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: G-10-20
Record Dates: First submitted 2020-11-08; First posted 2020-11-12 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Helicobacter Pylori Infection
Keywords: Doxycycline; LOAD regimen; Helicobacter Pylori; levofloxacine; tinadizole
MeSH Terms: interventions — Doxycycline; Esomeprazole; Ofloxacin; Levofloxacin; Amoxicillin; Omeprazole

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Doxycyclien (Experimental): Measure eradication rate of Helicobacter pylori infection with Doxycycline,Levofloxacien,tinadizole
  Interventions: Drug: Doxycycline
- Levofloxacine (Active Comparator): Measure eradication rate of Helicobacter pylori infection with Livofloxacine and tinadizole,amoxicilline
  Interventions: Drug: Levofloxacin 500mg

INTERVENTIONS:
Drug: Doxycycline — Doxycylcine 100 mg bid ,esomprazole 20 bid,levofloxacineq.d,Tinadizole 500 bid
  Other Names: Tinadizole; Esomeprazole; levofloxacine
  Arms: Doxycyclien
Drug: Levofloxacin 500mg — Levofloxacin 500 mg qd, amoxicillin 500 2cab bid,Tinadizole 500 bid, esomprazole 20 bid
  Other Names: Amoxicilline; Esomeprazol; Tinadizole
  Arms: Levofloxacine

SUMMARY:
Comparison Efficacy of two weeks Therapy with Doxycycline,levofloxacine,Tinadizole Versus Levofloxacine,Tinadizole,Amocillin on Eradication of Helicobacter Pylori in Syrian population.

ELIGIBILITY:
Inclusion Criteria:

* Patients are aged greater than 18 years old who have H. pylori infection diagnosed by any of following three methods:
* Positive rapid urease test (CLOtest).
* Histologic evidence of H. pylori by modified Giemsa staining.
* Positive 13C-urea breath test. without prior eradication therapy and are willing to receive therapy.

Exclusion Criteria:

* Children and teenagers aged less than 18 years.
* Previous eradication treatment for H. pylori.
* Patients who took any drug, which could influence the study results such as proton pump inhibitor, H2 blocker, mucosal protective agent and antibiotics.
* History of gastrectomy.
* Gastric malignancy, including adenocarcinoma and lymphoma,
* Previous allergic reaction to antibiotics (Amoxicillin, Tinadizole,
* Doxycycline,Bismuth subsalicylate,) and prompt pump inhibitors (Es- omeprazole).
* Contraindication to treatment drugs.
* Pregnant or lactating women.
* Severe concurrent disease.
* Liver cirrhosis.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-10-31 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
Eradication rate of Helicobacter pylori infection | 8 week from begning of treatment
  Eradication rate of Helicobacter infected patients

CONTACTS AND LOCATIONS:
Overall Officials: Marouf M Alhalabi, MD, Principal Investigator — general assambly of damascus hospital
Locations (1):
- General Assembly of Damascus Hospital, Damascus, Syria

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR
Time Frame: Within 5 year of study completion